CLINICAL TRIAL: NCT01650545
Title: A Pilot Study to Demonstrate Efficacy and Safety of Aerosol Liposomal Cyclosporine (L-CsA) in the Treatment of Bronchiolitis Obliterans Syndrome After Lung Transplantation
Brief Title: Aerosol Liposomal Cyclosporine for Chronic Rejection in Lung Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00049596
Record Dates: First submitted 2012-06-27; First posted 2012-07-26 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2018-03

CONDITIONS: Disorder Related to Lung Transplantation; Bronchiolitis Obliterans; Decreased Immunologic Activity; Chronic Rejection of Lung Transplant
Keywords: case-control study; aerosolized liposomal cyclosporine A; bronchiolitis obliterans syndrome; Lung Transplantation; Lung function
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome | interventions — Cyclosporine; Tacrolimus; Sirolimus

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Aerosol Cyclosporine (Experimental): Arm 1) Aerosol liposomal cyclosporine Open label randomized trial using experimental inhalational therapy with liposomal aerosol cyclosporine in addition to standard immune suppression (tacrolimus , mycophenolate mofetil and prednisone) for 6 month duration at inhalational doses (5mg and 10 mg bid), to be defined by transplant type respectively (single, double lung transplant )
  Interventions: Drug: Liposomal aerosol cyclosporine; Other: standard immune suppression, oral
- Conventional oral immune suppression (Active Comparator): Arm 2) Standard immune suppression consisting of typical oral immune suppression for lung transplant recipients typically tacrolimus, mycophenolate mofetil and prednisone.
  Conventrional oral immune suppression as standard of care thus consists of tacrolimus, mycophenolate mofetil prednisone rapamycin described in the subsequent section as well.
  Interventions: Other: standard immune suppression, oral

INTERVENTIONS:
Drug: Liposomal aerosol cyclosporine — inhaled form of immune suppression
  Other Names: cyclosporine
  Arms: Liposomal Aerosol Cyclosporine
Other: standard immune suppression, oral — conventional drug
  Conventrional oral immune suppression as standard of care thus consists of tacrolimus, mycophenolate mofetil prednisone and rapamycin
  Other Names: tacrolimus; rapamycin; sirolimus

SUMMARY:
This is a single-center pilot study to investigate the efficacy and safety of aerosolized liposomal cyclosporine A in the treatment of chronic rejection in lung transplant recipients with bronchiolitis obliterans syndrome (BOS).

The primary objective is to evaluate the efficacy of liposomal cyclosporine A in the treatment of chronic rejection. Pulmonary function and changes in BOS grade are the primary end points.

DETAILED DESCRIPTION:
This is a randomized single-center pilot study to investigate the efficacy and safety of aerosolized liposomal cyclosporine A (L-CsA) in the treatment of chronic rejection in lung transplant recipients with Grade 1 or 2 BOS.

The primary endpoints will include:

* Improvement or stabilization of pulmonary function test (FEV1) from baseline
* Stabilization of histology (no deterioration from baseline)
* Safety of the preparation

The secondary endpoints will include:

* Pharmacokinetics and distribution of CsA in blood -
* Change in cytokine levels from BAL specimens.

ELIGIBILITY:
Inclusion Criteria:

Chronic rejection

1. Bronchiolitis obliterans diagnosed by bronchiolitis obliterans syndrome and > 20% decline from the individual patient's best FEV1 is observed
2. Recipient of a double or single lung transplant
3. Receiving immunosuppressive treatment according to institutional standards

Exclusion criteria:

1. Active invasive bacterial, viral or fungal infection
2. Current mechanical ventilation
3. Pregnant or breast-feeding woman
4. Known hypersensitivity to cyclosporine A
5. Serum creatinine value of more than 265 μmol/L (3 mg/dL) or chronic dialysis
6. Receipt of an investigational drug as part of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo T Iacono, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Aerosol Cyclosporine: Arm 1) Aerosol liposomal cyclosporine Open label randomized trial using experimental inhalational therapy with liposomal aerosol cyclosporine in addition to standard immune suppression (tacrolimus , mycophenolate mofetil and prednisone) for 6 month duration at inhalational doses (5mg and 10 mg bid), to be defined by transplant type respectively (single, double lung transplant )
  Liposomal aerosol cyclosporine: inhaled form of immune suppression
  standard immune suppression, oral: conventional drug
- Conventional Oral Immune Suppression: Arm 2) Standard immune suppression consisting of typical oral immune suppression for lung transplant recipients typically tacrolimus, mycophenolate mofetil and prednisone
  standard immune suppression, oral: conventional drug
Period: Overall Study
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [35 to 81] | 63.8 [32 to 75] | 61.3 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Chronic Rejection Who Met Primary Combined End-point
Description: Treatment failure defined as: BOS progression (> 20% decline lung function), re-transplant, or death
Time Frame: approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression
Number analyzed (Participants) | 11 | 10
Participants | 2 | 5
Statistical Analysis 1: Comparison: Liposomal Aerosol Cyclosporine vs Conventional Oral Immune Suppression; Test type: Superiority; p = 0.03, Log Rank

2. Secondary Outcome: Cytokine Analysis From BAL Fluid in Lung
Description: Multiple cytokines were assessed as markers of lung inflammation that may be used in addition to biopsy data, collected per patient as clinically indicated during the follow-up interval. Values are reported as mean change from baseline in each group, per week
Time Frame: baseline to approximately 1 year
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression
Number analyzed (Participants) | 11 | 10
pg/mL
  lL-1beta | -2 [-9.3 to 5.3] | 3.3 [-4.3 to 10.9]
  IL-2 | -0.9 [-1.5 to 0.3] | -0.3 [-0.9 to 0.3]
  IL-6 | -2.0 [-7.9 to 3.9] | 6.3 [1.2 to 11.5]
  IL-8 | 13.6 [-20.3 to 47.4] | 37.5 [2.1 to 72.9]
  IL-10 | 0.1 [-0.7 to 0.9] | 0.1 [-1.3 to 1.5]
  IL-17 | 0.4 [-0.1 to 0.8] | 0.1 [-0.5 to 0.8]
  TNF-alpha | 1.9 [-8.6 to 12.4] | -1.7 [-8 to 4.7]
  IFN-gamma | 0.5 [-0.1 to 1] | 0 [-0.4 to 0.5]

3. Secondary Outcome: Overall Survival at 5 Years Follow-up
Description: Number of participants surviving at 5 year follow-up
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Liposomal Aerosol Cyclosporine: Arm 1) Aerosol liposomal cyclosporine Open label randomized trial using experimental inhalational therapy with liposomal aerosol cyclosporine in addition to standard immune suppression (tacrolimus , mycophenolate mofetil and prednisone) for 6 month duration at inhalational doses (5mg and 10 mg bid), to be defined by transplant type respectively (single, double lung transplant )
  Liposomal aerosol cyclosporine: inhaled form of immune suppression
  standard immune suppression, oral: conventional drug
  Conventrional oral immune suppression as standard of care thus consists of tacrolimus, mycophenolate mofetil prednisone and rapamycin
- Conventional Oral Immune Suppression: Arm 2) Standard immune suppression consisting of typical oral immune suppression for lung transplant recipients typically tacrolimus, mycophenolate mofetil and prednisone.
  Conventrional oral immune suppression as standard of care thus consists of tacrolimus, mycophenolate mofetil prednisone rapamycin described in the subsequent section as well.
  standard immune suppression, oral: conventional drug
  Conventrional oral immune suppression as standard of care thus consists of tacrolimus, mycophenolate mofetil prednisone and rapamycin
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression
Number analyzed (Participants) | 11 | 10
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events monitored for one year as described in the IND. All cause mortality monitored out to 5 years.
Arm/Group | Liposomal Aerosol Cyclosporine | Conventional Oral Immune Suppression
All-Cause Mortality (participants affected / at risk) | 6/11 | 10/10
Serious Adverse Events (participants affected / at risk) | 8/11 | 8/10
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Aerosol Cyclosporine (N=11) | Conventional Oral Immune Suppression (N=10)
Atrial flutter (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Rapid atrial fibrillation (Cardiac disorders) | 0 | 1
Cholelithiasis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 0 | 2
Weakness (General disorders) | 0 | 1
Acute graft rejection (Immune system disorders) | 3 | 1
Bacteremia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Herpes zoster exacerbation (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 4
Pyrexia (Infections and infestations) | 0 | 1
Respiratory syncytial virus (Infections and infestations) | 0 | 3
Rhinovirus (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Squamous cell carcinoma (scalp/left cheek) (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Aerosol Cyclosporine (N=11) | Conventional Oral Immune Suppression (N=10)
Atrial flutter (Cardiac disorders) | 1 | 0
Carotid atherosclerosis (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Rapid atrial fibrillation (Cardiac disorders) | 0 | 1
Ear inflammation (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 2 | 1
Cholelithiasis (Gastrointestinal disorders) | 1 | 0
Clostridium difficile (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Emesis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 2
Allergic rhinitis (General disorders) | 0 | 1
Ankle edema (General disorders) | 1 | 1
Ankle pain (General disorders) | 1 | 0
Back pain (General disorders) | 3 | 3
Bilateral ankle edema (General disorders) | 1 | 1
Bilateral foot edema (General disorders) | 1 | 2
Bilateral knee pain (General disorders) | 0 | 1
Bilateral leg edema (General disorders) | 1 | 2
Elevated creatinine level (General disorders) | 1 | 0
Elevated tacrolimus level (General disorders) | 1 | 0
Fall (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Generalized pain (in joints) (General disorders) | 1 | 0
Left knee pain (General disorders) | 1 | 0
Leg edema (General disorders) | 1 | 0
Low back pain (General disorders) | 3 | 0
Malaise (General disorders) | 6 | 1
Motor vehicle crash (General disorders) | 1 | 0
Muscle spasms (General disorders) | 1 | 0
Neck edema (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Paresthesia (lower legs) (General disorders) | 0 | 2
Right leg weakness (General disorders) | 0 | 1
Shoulder and back pain (General disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cytomegalovirus (Infections and infestations) | 1 | 0
Herpes zoster exacerbation (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Lower respiratory infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 5
Pyrexia (Infections and infestations) | 1 | 1
Respiratory syncytial virus (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 1 | 1
Rhinovirus (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Confusion (Nervous system disorders) | 1 | 0
Hallucinations (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Uterine pain (Reproductive system and breast disorders) | 0 | 1
Acute rejection (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspepsia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Abscess (right axillary) (Skin and subcutaneous tissue disorders) | 1 | 0
Anterior tongue lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Foot rash (Skin and subcutaneous tissue disorders) | 1 | 0
Herpes zoster (left scalp, ear, face) (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1
Squamous cell carcinoma (chest, temple) (Skin and subcutaneous tissue disorders) | 1 | 0
Squamous cell carcinoma (scalp/left cheek) (Skin and subcutaneous tissue disorders) | 1 | 0
Squamous cell carcinoma (left ear) (Skin and subcutaneous tissue disorders) | 0 | 1
Squamous cell carcinoma (left hand) (Skin and subcutaneous tissue disorders) | 0 | 1
Urticarial (left cheek) (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Postural hypotension (Vascular disorders) | 0 | 1
Pulmonary hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No